CLINICAL TRIAL: NCT03274284
Title: Chemoradiotherapy for Recurrent T1G3 Bladder Cancer After BCG Failure
Brief Title: Chemoradiotherapy for Recurrent T1G3 Bladder Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MokhtarDawood, Assistant Lecturer of Urology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bl Cancer
Record Dates: First submitted 2017-08-29; First posted 2017-09-06 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Bladder Cancer
Keywords: chemoradiation for; T1G3 BC
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemoradiotherapy (Experimental): Chemoradiation in the form of cisplatin plus conformal radiotherapy 55GY/20 fractions which is biologically effective to 64GY/32 fractions fr
  Interventions: Combination Product: chemoradiation

INTERVENTIONS:
Combination Product: chemoradiation — chemoradiation in case of T1G3 BC after BCG failure.

SUMMARY:
To evaluate the short term results of chemoradiation in case of T1G3 BC after BCG failure.

DETAILED DESCRIPTION:
Non- muscle invasive bladder cancer (NMIBC) is a heterogeneous group of cancers. For most urologists the treatment of T1G3 tumor poses a dilemma of management.The spectrum of clinical behavior includes; T1 lesions that will not progress however T1G3 may be potentially lethal, associated with metastatic disease at the time of presentation.

The major goal of treatment for T1G3 BC should be bladder preservation whenever possible.

Intravesical therapy with Bacille Calmette Guerin (BCG) may decrease the recurrence rate by compared with transurethral resection of bladder tumor (TURBT) alone.

ELIGIBILITY:
Inclusion Criteria:

* All patients with recurrent T1G3 bladder cancer after 6 doses of BCG consenting for chemoradiation and refusing radical cystectomy

Exclusion Criteria:

* Any patients with distant metastasis or positive LN on CT or MRI.
* Patients unfit for chemoradiation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Result of chemoradiation for recurrentT1G3 BC after BCG failure | followup within two years
  treatment of 20 patients with recurrent T1G3
  BC by chemoradiation to see efficacy and safety .and to reduce the number of recurrent cases and improve survival.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Moeen, Study Director — Moeen3@yahoo.com

REFERENCES:
- [Background] Lambert EH, Pierorazio PM, Olsson CA, Benson MC, McKiernan JM, Poon S. The increasing use of intravesical therapies for stage T1 bladder cancer coincides with decreasing survival after cystectomy. BJU Int. 2007 Jul;100(1):33-6. doi: 10.1111/j.1464-410X.2007.06912.x. PMID 17552951
- [Background] Soloway MS, Sofer M, Vaidya A. Contemporary management of stage T1 transitional cell carcinoma of the bladder. J Urol. 2002 Apr;167(4):1573-83. PMID 11912367